CLINICAL TRIAL: NCT06613893
Title: Effect of Inhalational Anesthesia Versus Total Intravenous Anesthesia on Blood Glucose Level in Type 2 Diabetes Mellitus Patients Undergoing Thoracic Surgery : a Comparative Study
Brief Title: Effect of Inhalational Anesthesia Versus Total Intravenous Anesthesia on Blood Glucose in Type 2 Diabetes Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Yasser Alaa Abdalmonim, Principal Investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: FMASU@MD331/2023
Record Dates: First submitted 2024-09-06; First posted 2024-09-26 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Type 2 Diabetes Mellitus (T2DM); Thoracic Surgery
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Fentanyl; Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A will receive total inravenous anesthesia (TIVA) (Active Comparator): patients in this group will receive total intravenous anesthesia using propofol infusion after induction of anesthesia, tested variables will be measured according to the protocol
- Group B will receive inhalational anesthesia (IHA) (Active Comparator): patients in this group will receive inhalational anesthesia using isoflurane, tested variables will be measured according to the protocol
  Interventions: Drug: Inhalational anesthesia

INTERVENTIONS:
Drug: TIVA — Anesthesia will be maintained by total intravenous anesthesia with propofol infusion (4 to 12 mcg/kg/min) and fentanyl infusion (1-2mcg /kg/hour) that will be stopped 30 min before the end of the operation ,The heart rate and blood pressure will be maintained within the range of ±20% of the baseline
  Other Names: Fentanyl; propofol
Drug: Inhalational anesthesia — Anesthesia will be maintained with inhaled isoflurane, Iso-MAC from (0.7 to 1.4%)(Hawkley, Preston, and Maani 2018) and fentanyl infusion (1-2mcg /kg/hour) that will be stopped 30 min before the end of the operation ,The heart rate and blood pressure will be maintained within the range of ±20% of the baseline
  Arms: Group B will receive inhalational anesthesia (IHA)

SUMMARY:
The aim of this study is to compare the effect of total intravenous anesthesia (TIVA) and inhalational anesthesia (IHA) as maintenance anesthesia on blood glucose level and complications in type 2 diabetic patients undergoing thoracic surgery . All participants had to understand and give written informed consent , and ethical committee approval (of Faculty of Medicine, Ain Shams University) will be obtained before participants allocation.

DETAILED DESCRIPTION:
* Type of Study: prospective , randomized .
* Study Settings: Ain Shams University hospitals, Cairo, Egypt.
* Study period: 12 months starting from janurary 2024 .
* Study Population: All adult type 2 diabetic patients (30-70 year old) with class II,III based on the American Society of Anesthesiologists (ASA) physical status undergoing elective thoracic surgeries will be randomly assigned into one of the following groups using computer generated codes and opaque sealed envelopes:

  1. Group A will receive total inravenous anesthesia (TIVA).
  2. Group B will receive inhalational anesthesia (IHA)

ELIGIBILITY:
Inclusion Criteria:

* Age 30 - 70 years
* Sex: Both sexes
* Patients with type 2 diabetes mellitus controlled with oral hypoglycemic drugs
* Patients with ASA classification II,III
* Duration of surgery (≥2 h)

Exclusion Criteria:

* Declining to give written informed consent
* ASA classification Ⅳ to V
* Severe systemic diseases
* Metabolic disorders, diabetic ketoacidosis or hyperglycemia (fasting blood Glucose more than 140 mg/dl)
* Hepatic and/or renal dysfunction
* Neuromuscular disease
* Pancreatic cancer
* History of malignant hyperthermia
* Emergency surgery
* Ischemic heart disease and valvular heart disease
* Body mass index more than 40
* Diabetic patients on insulin therapy

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Blood glucose levels in milligrams per decilitre (mg/dl) at different time points | Immediate preoperative till 48 hours after recovery from anesthesia
  Blood glucose levels in milligrams per deciliter at different time points: preoperative (T0), post-intubation (T1), 1st , 2nd and 3rd hour after the start of the operation (T3, T4 and T5, respectively), 1st hour after the operation (T6) , 2nd hour after the operation (T7), 1st and 2nd day after the operation (T8, T9)

SECONDARY OUTCOMES:
Serum insulin level in picomoles per litre (pmol/l) | 30 min before induction of anesthesia and 30 min after surgery and recovery from anesthesia
  serum insulin level (pmol/l) 30 min before and 30 min after surgery
Serum cortisol level in micrograms per decilitre (mcg/dl) | 30 min before induction of anesthesia and 30 min after surgery and recovery from anesthesia
  serum cortisol level (mcg/dl) 30 min before and 30 min after surgery
The incidence of postoperative complications | The complications will be assessed on the first, third and seveth post-operative day
  The complications that will be tested Acute coronary syndrome. Stroke. acute kidney injury. stress gastric ulcer. surgical site infection. Hypoglycaemia (blood glucose level below 70 mg/dL). Hyperglycemia (fasting blood glucose level greater than 125mg/dL while 2 hours postprandial greater than 200 mg/dL).
  Postoperative nausea and vomiting . postoperative pulmonary complications including atelectasis, pneumonia and respiratory failure

CONTACTS AND LOCATIONS:
Overall Officials: Nabila M Abdelaziz, professor, Study Director — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No